CLINICAL TRIAL: NCT00852267
Title: Lipoprotein Effects of Substituting Beef Protein for Carbohydrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2007-068
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Healthy; Cardiovascular Disease; Atherogenic Dyslipidemia
Keywords: cholesterol; diet; protein; carbohydrate; saturated fat; LDL subclass; healthy volunteers
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- High CHO, High SatFat Diet (Active Comparator)
  Interventions: Other: High Carbohydrate, High Saturated Fat Diet
- Low CHO, High SatFat Diet (Experimental)
  Interventions: Other: Low Carbohydrate, High Saturated Fat Diet
- Low CHO, Low SatFat Diet (Experimental)
  Interventions: Other: Low Carbohydrate, Low Saturated Fat Diet

INTERVENTIONS:
Other: High Carbohydrate, High Saturated Fat Diet — 50% Carbohydrate; 12% Protein; 38% Fat (15% Saturated Fat; 15% Monounsaturated Fat)
  Arms: High CHO, High SatFat Diet
Other: Low Carbohydrate, High Saturated Fat Diet — 31% Carbohydrate; 31% Protein; 38% Fat (15% Saturated Fat; 14% Monounsaturated Fat)
  Arms: Low CHO, High SatFat Diet
Other: Low Carbohydrate, Low Saturated Fat Diet — 31% Carbohydrate; 31% Protein; 38% Fat (8% Saturated Fat; 21% Monounsaturated Fat)
  Arms: Low CHO, Low SatFat Diet

SUMMARY:
The purpose of this study is to test whether replacing dietary carbohydrate with protein, using beef as the primarily source of protein, will improve risk factors for cardiovascular disease.

DETAILED DESCRIPTION:
The primary aim of this study is to test the hypothesis that replacing dietary carbohydrate with protein, using beef as the primarily source of protein, will have beneficial effects on components of atherogenic dyslipidemia and postprandial lipoprotein response and that these effects will be independent of saturated fat intake.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure less than 150/90
* Body mass index (BMI)≥ 20 and ≤ 35 kg/m2
* Non-smoker
* Agrees not to consume alcohol during the study
* Agrees to abstain from taking dietary supplements during the study
* LDL-cholesterol and total cholesterol < 95th percentile for age and sex
* Fasting triglycerides < 500 mg/dL
* Fasting glucose concentration < 126 mg/dL
* Hematocrit (HCT) ≥ 36%
* At least three months of a weight-stable state (± 3% of body weight)

Exclusion Criteria:

* Personal history of coronary heart disease, cerebrovascular disease, peripheral vascular disease, diabetes, lung disease, bleeding disorder, liver or renal disease, HIV or of cancer (other than skin cancer) in the last five years
* Taking drugs known to affect lipid metabolism or insulin resistance, hormones, or the blood thinning agent warfarin
* Abnormal thyroid stimulating hormone (TSH)
* Strength trains with resistance weights more than four hours per week

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | 3 weeks, 8 weeks, and 13 weeks
Non-HDL Cholesterol | 3 weeks, 8 weeks, and 13 weeks
Apolipoprotein B | 3 weeks, 8 weeks, and 13 weeks
LDL-Cholesterol/HDL-Cholesterol | 3 weeks, 8 weeks, and 13 weeks
Apolipoprotein B/Apolipoprotein AI | 3 weeks, 8 weeks, and 13 weeks

SECONDARY OUTCOMES:
LDL peak diameter | 3 weeks, 8 weeks, and 13 weeks
LDL subclass 3 (LDL3) | 3 weeks, 8 weeks, and 13 weeks
HDL subclass 2 (HDL2) | 3 weeks, 8 weeks, and 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States

REFERENCES:
- [Derived] Mangravite LM, Chiu S, Wojnoonski K, Rawlings RS, Bergeron N, Krauss RM. Changes in atherogenic dyslipidemia induced by carbohydrate restriction in men are dependent on dietary protein source. J Nutr. 2011 Dec;141(12):2180-5. doi: 10.3945/jn.111.139477. Epub 2011 Oct 26. PMID 22031660